CLINICAL TRIAL: NCT06733441
Title: Phase 1b, Randomized, Dose Optimization Study to Assess the Anti-Tumor Activity, Safety, and Pharmacokinetics of TLN-254 in Patients With Relapsed or Refractory T-cell Lymphoma
Brief Title: A Study of TLN-254 in Participants With Relapsed or Refractory T-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Treeline Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLN-254-2401
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma
Keywords: Relapsed or refractory Cutaneous T Cell Lymphoma; Relapsed or refractory Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence; Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: TLN-254 Single Agent (Experimental)
  Interventions: Drug: TLN-254
- Cohort 2: TLN-254 Single Agent (Experimental)
  Interventions: Drug: TLN-254

INTERVENTIONS:
Drug: TLN-254 — TLN-254 will be administered orally at a specified dose on specified days depending on treatment allocation.
  Arms: Cohort 1: TLN-254 Single Agent
Drug: TLN-254 — TLN-254 will be administered orally at a specified dose on specified days.
  Arms: Cohort 2: TLN-254 Single Agent

SUMMARY:
The primary purpose of this study is to evaluate the anti-tumor activity of TLN-254 monotherapy in participants with relapsed or refractory T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Age:

1. At least 18 years of age at the time of signing the informed consent form (ICF).

   Type of Participant and Disease Characteristics:
2. Cohort 1: Peripheral T-cell lymphoma (PTCL) that has relapsed after, or not responded to at least one prior systemic treatment regimen. Participants with Anaplastic large cell lymphoma (ALCL) should have received prior brentuximab vedotin treatment.

   * Nodal T-follicular helper (TFH) cell lymphoma angioimmunoblastic; Follicular helper T-cell lymphoma, angioimmunoblastic type (angioimmunoblastic T-cell lymphoma).
   * Nodal TFH cell lymphoma, follicular type; Follicular helper T-cell lymphoma, follicular type.
   * Nodal TFH cell lymphoma, not otherwise specified (NOS); Follicular helper T-cell lymphoma, NOS.
   * PTCL, NOS.
   * Anaplastic large-cell lymphoma, Alkaline phosphatase (ALK) positive.
   * Anaplastic large-cell lymphoma, ALK negative.

   Cohort 2: Relapsed/refractory CTCL which has relapsed after, or not responded to at least two prior systemic treatments.
   * Sezary syndrome
   * Mycosis fungoides
3. Participant must have measurable disease at study entry.
4. Freshly biopsied or archival tissue available.

   Diagnostic Assessments:
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
6. Adequate organ function.

   Contraception:
7. Participants must accept and follow the pregnancy prevention plan.

Exclusion Criteria:

Medical Conditions:

1. Participants must not have prior systemic anti-cancer treatment less than or equal to (≤) 5 half-lives or 4 weeks, allogeneic SCT≤90 days or autologous SCT ≤60 days prior to study intervention initiation.
2. Participants must not have any condition, including significant acute or chronic medical illness, active or uncontrolled infection, or the presence of laboratory abnormalities, that places participants at unacceptable risk if participating in this study.
3. Current or past history of central nervous system (CNS) involvement.

Other Exclusions:

* Pregnant or lactating women.
* Unable to swallow tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response | Up to 2 years
Percentage of Participants With CR | Up to 2 years
Percentage of Participants With PR | Up to 2 years

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 2 years
Number of Participants With Severity of TEAEs Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 | Up to 2 years
Plasma concentrations of TLN-254 | Day 1 of Cycle 1 and Day 1 of each even numbered Cycle for up to 2 years (Each Cycle length =28 days)
Duration of Response (DOR) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Stanford Cancer Institute, Stanford, California
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No